CLINICAL TRIAL: NCT02920333
Title: Efficacy of the Non-invasive Brain Stimulation Techniques for Lower Limb Recovery in Stroke Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The grant funding has expired
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIBS2014/00359
Record Dates: First submitted 2014-12-21; First posted 2016-09-30 (Estimated); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Stroke
Keywords: stroke; transcraniel direct current stimulation; repetitive transcraniel magnetic stimulation; rehabilitation; lower extremities
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- tDCS+ rehab training (Experimental): tDCS will be applied 10 days, followed by conventional rehab training. Anodal stimulation will be conducted at the intensity of 2 mA and last for 20 minutes over the affected primary motor cortex of cortical representation of the tibialis anterior muscle.
  Interventions: Procedure: conventional rehab training; Device: tDCS
- rTMS+ rehab training (Experimental): rTMS will be applied 10 days, followed by conventional rehab training. Subjects will receive 10 Hz rTMS, and a total of 1200 pulses will be delivered for one treatment session.
  Interventions: Procedure: conventional rehab training; Device: rTMS
- sham tDCS+ rehab training (Sham Comparator): The same stimulation parameters as tDCS treatment will be employed for the sham stimulation. However, the current will be applied for 30 seconds only, to give subjects the sensation of the stimulation.
  Interventions: Procedure: conventional rehab training; Device: sham tDCS

INTERVENTIONS:
Procedure: conventional rehab training — Conventional rehab training will be conducted daily for 10 days, after NIBS intervention.
Device: tDCS — tDCS will be applied 10 days, followed by conventional rehab training. Stimulation will be conducted at the intensity of 2 mA and last for 20 minutes. anode will be placed over the affected primary motor cortex (M1) of cortical representation of the tibialis anterior muscle (TA), while the cathode will be used as reference electrode and placed over the forehead of the unaffected side.
  Arms: tDCS+ rehab training
Device: rTMS — rTMS will be applied 10 days, followed by conventional rehab training. Subjects will receive 10 Hz rTMS, and a total of 1200 pulses will be delivered for one treatment session.
  Arms: rTMS+ rehab training
Device: sham tDCS — The same stimulation parameters as tDCS treatment will be employed for the sham stimulation. However, the current will be applied for 30 seconds only, to give subjects the sensation of the stimulation.
  Arms: sham tDCS+ rehab training

SUMMARY:
This study is to compare the efficacy of two types of non-invasive brain stimulation (NIBS) in lower limb motor function recovery in stroke patients. The intervention will be tDCS (transcraniel direct current stimulation) or rTMS (repetitive transcraniel magnetic stimulation) plus conventional gait training for 10 days over 2 weeks.

The study hypothesizes that:

1. When combined with conventional gait training, NIBS could improve the walking ability of stroke survivors.
2. NIBS will modulate cortex activity of the brain area representing the lower limbs.
3. The effects of NIBS might be related to some genetic factors. 45 subjects will be randomly divided into 3 groups, receiving tDCS plus conventional gait training, or rTMS plus conventional gait training, or sham tDCS plus conventional gait training.

The outcome measures include clinical functional assessment, brain activity assessed by TMS measurement and MRI, genetic factor measurement. All these will be done at pre, immediate after intervention and 4 weeks after intervention.

DETAILED DESCRIPTION:
This is an exploratory randomized trial on 45 subacute stroke subjects with gait impairment following a single anterior circulation subcortical stroke 3-6 months prior to recruitment, with comfortable walking speed of 0.2 to 0.4 m/s (which generally describes those who require 1 person assistance to supervision for ambulation - Functional Ambulatory Category (FAC) 3 (Kollen, et al. 2006). Exclusion criteria include a history of seizures, uncontrolled medical condition or psychiatric history, neglect, aphasia, or any cognitive or behavioural impairment causing inability to comply with instructions, cranial surgeries, pacemakers and other implants which preclude the use of NIBS. Subjects on psychoactive medications (eg. antiepileptics, antipsychotic and antidepressant medications) will be excluded from the study. The diagnosis for subjects' eligibility to join the study will be determined by subjects' self-report (to obtain medical history), medical records (to verify subjects' self-report) as well as assessment by the research staff in the screening session (including FMA and 10 meter walk test, ). Subjects should have completed inpatient rehabilitation and should not be undergoing any other interventions targeting lower limb recovery during the study. Subjects are allowed to continue with outpatient rehabilitation (generally not more than twice a week) and home exercise program after the active intervention phase of the study.

45 subjects with stroke will be recruited and randomized into 3 groups by a randomization stratification approach with a computer-generated random sequence. Group 1 to receive facilitatory 2 mA anodal tDCS for 20min to the affected M1 motor cortical representation of the tibialis anterior muscle (TA) together with conventional post-stroke functional mobility training; Group 2 to receive 2000 pulses of 10 Hz facilitatory rTMS to the affected motor cortex with conventional therapy; Group 3 to receive sham stimulation with conventional therapy. All groups will receive 2 weeks (10 days) of tDCS, rTMS or sham stimulation combined with daily standardized post-stroke conventional training in functional mobility.

tDCS A research staff supervised by a physician will apply the tDCS to the subject. Direct current will be transferred by a saline-soaked pair of surface sponge electrode (35cm2) and delivered by a battery-operated, constant current stimulator with a maximum output of 10mA, through a non-metallic conductor rubber electrode. Stimulation will be conducted at the intensity of 2 mA and last for 20 minutes. The anode will be placed over the affected primary motor cortex (M1) of cortical representation of the tibialis anterior muscle (TA), while the cathode will be used as reference electrode and placed over the forehead of the unaffected side.

Sham stimulation The same stimulation parameters as tDCS treatment will be employed for the sham stimulation. However, the current will be applied for 30 seconds only, to give subjects the sensation of the stimulation. This method of sham stimulation has also been validated (Gandiga et al., 2006). Current intensity will be increased and decreased gradually to decrease perception rTMS A research staff supervised by a physician will apply the intervention of rTMS to the subject. For all TMS procedures, patients will be seated comfortably and instructed to remain as still as they can. The height of the chair will be adjusted so that both the knees and ankles are flexed at 90 degree and the two feet rest on the floor. A tight swim cap will be worn by the subject. The vertex will be marked on the cap. Points that are 1 cm lateral and/or 1cm posterior/anterior are marked on the cap.

Subjects will receive 10 Hz rTMS using Magstim Rapid2, with the double cone coil placed over the "hot spot" of the affected M1. The stimulation intensity will set as 90% of RMT (or 80% AMT, if RMT is not available), and a total of 2000 pulses will be delivered for one treatment session.

Outcome measures will be obtained before, after the 2-week intervention and 4 weeks post-intervention, and will include 1) clinical measures (FAC, gait analysis, 10 meter walk test, 6 minute walk test, timed up and go), 2) cortical excitability measures using TMS (changes in resting motor threshold (RMT), or active motor threshold (AMT) of the affected and unaffected TA and short-interval cortical inhibition/facilitation (SICI/SICF), measured according to the technique of Rossini et al. (1994)), 3) MRI measures including diffusion tensor tractography (DTT), resting state protocols and GABA scan. 4) Genotyping and blood level of BDNF. 5) Psychological and cognitive assessment including Beck Depression Inventory (BDI), Fatigue Severity Scale, forward and backward digit span.

Clinical measures (10 meter walk test, 6 minute walk test, timed up-and-go test, gait analysis) A research staff supervised by a physical therapist will perform the functional assessment to the subject at the National University Hospital. The functional assessment consists of a 10 meter walk test, 6 minute walk test and a timed up-and-go test performed in a randomized order. The tester will not provide any assistance as the patient makes their way around the track, however, the tester will shadow the patient so as to attend to any problems should there be a need to.

The 10 meter walk test will be performed in a quiet indoor track of 14 meters long. Subject should walk at his comfortable pace as usual. The test will be repeated 3 times and the average of the duration to finish the 10 meter walk and total steps will be recorded.

The 6-minute walking test will be performed in an indoor track marked at 5-metre intervals. Subject should walk at his comfortable pace as usual. The distance over 6 minutes will be measured.

The timed up-and-go test will involve the subject getting off a standard armchair from a seated position, walking 3 meters from the chair, turning back and walking to the chair and seating back down. Subject should walk at his comfortable pace as usual. The test will be repeated 3 times and the duration the subject takes to perform the whole task will be recorded and averaged.

10 meter walk test, 6 minute walk test, timed up-and-go test altogether will take around 30 minutes, including set-up time.

Gait analysis will be performed using the Tekscan walkway system. Subjects will be required to walk on a mat at their comfort speed and the process might be video-recorded for future analyzing the quality of subjects' movement (face will not be captured and consent will be obtained in advance). Gait parameters including step and stride parameters, symmetry scores, velocity, and cadence temporal will be collected and recorded while the subject is walk along the walkway. The whole procedure will last up to 30 minutes.

TMS A research staff supervised by a physician will apply the TMS measurement of the cortical excitability and intracortical inhibition/facilitation to the subject. For all TMS procedures, patients will be seated comfortably and instructed to remain as still as they can. The height of the chair will be adjusted so that both the knees and ankles are flexed at 90 degree and the two feet rest on the floor. A tight swim cap will be worn by the subject. The vertex will be marked on the cap. Points that are 1 cm lateral and/or 1cm posterior/anterior are marked on the cap.

Single pulse TMS-Resting motor threshold (RMT) measurement Singe pulse TMS was delivered using Magstim Bistim² stimulator via a double cone coil. The double cone coil was oriented to induce a posterior-anterior current flow in cortex. The coil was placed on the cap with the intersection of the two embedded coils located over the marked point. The coil position was maintained manually by an assistant. Surface electromyography (EMG) electrodes are attached to the TA for EMG recording. The "hot spot" of the motor evoked potential (MEP) from TA is identified first from one of the marked points for both left and right side. This spot was marked on the elastic cap and used for all recordings on that side. The lowest intensity needed to elicit a MEP response of at least 50µV amplitude and that has been elicited in 50% of 8 successive trials will be recorded as RMT.

Single pulse TMS-Active motor threshold (AMT) The measurement of AMT is similar with RMT measurement. Except that subject's feet were constrained by flexible weights placed over the dorsum of each foot to ensure isometric activation. The subject was given real time feedback of EMG on an oscilloscope to match a target contraction corresponding to 20% maximal voluntary isometric contractions (MVIC) for TA. The lowest intensity needed to elicit a MEP response of at least 100µV amplitude at the "hot spot" and that has been elicited in 50% of 8 successive trials will be recorded as AMT.

Paired-pulse TMS- intracortical inhibition/facilitation measurement A first subthreshold conditioning stimulus (80% of RMT) will be applied, followed by a second suprathreshold stimulus (120% of RMT) with a variable interstimulus interval (ISI). The following ISIs - 2, 3, 4, 6, 9, 10, 12, 15 ms will be used. The percentage of change for each ISI before and after TMS will be calculated from the MEPs and will therefore provide a measure of change in intracortical facilitation and inhibition. Both single- and paired-pulse paradigms will be performed on the affected and unaffected hemisphere.

MRI scan (resting MRI, DTI scan [diffusion tensor Imaging], GABA scan) MRI scan will be performed at CIRC, NUS by the staff of CIRC. Prior to the scan, all subjects will be briefed of the test procedure and safety aspects. All participants will be scanned on a 3-T GE scanner using a standard radiofrequency head coil. Head motion was minimized by foam padding and forehead-restraining straps.

Psychological and cognitive assessment A research staff will conduct Beck Depression Inventory (BDI), Fatigue Severity Scale, forward and backward digit span. Digit Span is neuropsychological test widely used to assess executive abilities following stroke and is sensitive to brain damage (Tamez et al., 2011). The Beck's Depression Inventory will be used to screen for major depression. As tDCS has been investigated for use in the treatment of depression and cognitive impairment, we added the digit span to control for confounding effect of cognitive improvement in this study.For subjects who screen positive for major depression or suicidal ideation, the investigator performing the screening will inform a physician investigator who will assess and make the necessary referral for psychiatric assessment and management.

Blood BDNF level measurement and Genotyping of BDNF Blood will be taken by a trained research staff/research nurse and analyzed at Neuroscience Laboratory, located at the Translational Medicine Centre, Yong Loo Lin School using in-house and commercial assays. 10-20 ml of blood will be taken each time via venipuncture for three times, at before intervention, after and 4 weeks after intervention, respectively, that is, at the same time point of other outcome measurement. In total, 30-60 ml of blood will be collected for each subject for the whole research study. 10ml of blood will be taken from 5 healthy subjects as controls which is needed by the BDNF analysis protocol. To minimize the laboratory error during the test procedure, each blood sample will be processed first to extract plasma and plasma will be stored at -80°C at Tissue Repository, NUH, until all blood samples are collected. All plasma samples will be analysed together after the last collection of blood from the last subject. Any blood specimens obtained during the study will be stored and analyzed only for the purposes of this study for a period not exceeding 5 years and will be destroyed after completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* For subjects receiving intervention:

  1. Male or female aged 21-80 years;
  2. First ever haemorrhagic or ischaemic subcortical stroke of 3-6 months prior to study enrolment;
  3. Functional Ambulatory Category 3 (requires not more than minimal assistance for walking);
  4. Be able to provide informed consent.
* For healthy subjects:

  1. Male or female aged 21-80 years;
  2. Physically healthy;
  3. Be able to provide informed consent.

Exclusion criteria:

* For subjects receiving intervention:

  1. Severe claustrophobia;
  2. pregnancy;
  3. cardiac pacemakers;
  4. orthodontics (braces);
  5. metal implant;
  6. presence of other non MRI-compatible ferromagnetic implants;
  7. history of epilepsy;
  8. sensorimotor disturbance due to other causes other than stroke;
  9. severe pain in the lower limbs affecting gait;
  10. uncontrolled medical conditions including hypertension, diabetes mellitus and unstable angina;
  11. major depression and a history of psychotic disorders (Subject with BDI score more than 30 will be excluded).
* For healthy subjects:

  1. Cardiovascular diseases;
  2. Diabetes mellitus;
  3. Pulmonary diseases;
  4. Smoker.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
changes of " gait parameters" from baseline to post-intervention and 4 weeks after intervention | before intervention, immediately after intervention, 4 weeks after intervention
  Gait analysis will be performed using the Tekscan walkway system. Subjects will be required to walk on a mat at their comfort speed. Gait parameters including step and stride parameters, symmetry scores, velocity, and cadence temporal will be collected and recorded while the subject is walking along the walkway.

SECONDARY OUTCOMES:
changes of "cortical excitability measured by TMS" from baseline to post-intervention and 4 weeks after intervention | before intervention, immediately after intervention, 4 weeks after intervention
  Subjects will be seated comfortably with both knees and ankles flexed at 90 degree and the two feet resting on the floor. A tight swim cap will be worn by the subject, the proposed stimulation sites will be marked on the cap. Magstim Bistim² stimulator and a double cone magnetic coil will be used for the TMS assessment. Resting motor threshold (RMT) or Active motor threshold (AMT), and intracortical inhibition/facilitation will be measured for the motor cortex representing tibialis anterior muscle in both hemisphere.
changes of " Blood BDNF level" from baseline to post-intervention and 4 weeks after intervention | before intervention, immediately after intervention, 4 weeks after intervention
  10-20 ml of blood will be taken each time via venipuncture for three times.
changes of " cortical excitability measured by fMRI" from baseline to post-intervention and 4 weeks after intervention | before intervention, immediately after intervention, 4 weeks after intervention
  MRI scan will be performed at CIRC, NUS by the staff of CIRC. Prior to the scan, all subjects will be briefed of the test procedure and safety aspects. All participants will be scanned on a 3-T GE scanner using a standard radiofrequency head coil. Head motion was minimized by foam padding and forehead-restraining straps.
changes of " Psychological and cognitive properties" from baseline to post-intervention and 4 weeks after intervention | before intervention, immediately after intervention, 4 weeks after intervention
  Beck Depression Inventory Fatigue Severity Scale Forward and backward digit span
changes of walking speed measured by "10 meter walk test" from baseline to post-intervention and 4 weeks after intervention | before intervention, immediately after intervention, 4 weeks after intervention
  The 10 meter walk test is a test of walking speed.
changes of walking distance measured by "6 minute walk test " from baseline to post-intervention and 4 weeks after intervention | before intervention, immediately after intervention, 4 weeks after intervention
  The 6-minute walking test will be performed in an indoor track marked at 5-metre intervals. Subject should walk at his comfortable pace as usual. The distance over 6 minutes will be measured.
changes of " timed up-to-go test " from baseline to post-intervention and 4 weeks after intervention | before intervention, immediately after intervention, 4 weeks after intervention
  The timed up-and-go test is a measurement of mobility. It includes a number of tasks such as standing from a seating position, walking, stopping, and sitting down. For the test, the person is asked to stand up from a standard chair and walk a distance of approximately 3 around and walk back to the chair and sit down again.

CONTACTS AND LOCATIONS:
Overall Officials: Effie Chew, MD, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore